CLINICAL TRIAL: NCT06635239
Title: Massive Open Online Course for Women with Breast Cancer: Development and Evaluation of an Intervention on Person-Centered Care and Digital Health Literacy in Breast Cancer
Brief Title: Massive Open Online Course (MOOC) for Women with Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yolanda Alvarez-Perez (Other)
Collaborators: Servicio de Evaluación del Servicio Canario de Salud (Unknown); Fundacion Canaria Instituto de Investigacion Sanitaria de Canarias (Other); University of La Laguna (Other); University of Barcelona (Other); FEFOC fundation (Unknown); Parc Taulí Hospital Universitari (Other); Hospital Clinic of Barcelona (Other); Universitat Autonoma de Barcelona (Other)
Responsible Party: Sponsor-Investigator, Yolanda Alvarez-Perez, PhD, Servicio Canario de Salud
Organization: Servicio Canario de Salud (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PIFIISC 19/24; CHUNSC_2019_61 (Other: Ethics Committee of Hospital Universitario Nuestra Señora de la Candelaria)
Record Dates: First submitted 2024-10-04; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: Massive Open Online Course; Digital Health Literacy; Health Literacy; Person-Centered Care
MeSH Terms: conditions — Breast Neoplasms | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-arm intervention (Experimental): Co-creation with women with breast cancer, their families, and healthcare professionals of a MOOC aimed at women with breast cancer; and evaluation of the MOOC's effectiveness and acceptability.
  Interventions: Other: Co-creation and assessment

INTERVENTIONS:
Other: Co-creation and assessment — 1. MOOC co-creation: development of a MOOC initially structured into modules consisting of a variety of downloadable educational resources such as videos, audios, infographics, texts, etc., covering several units related to Person-Centered Care (Shared Decision-Making, strategies for managing the clinical encounter, Patient Decision Aids, etc.) and Digital Health Literacy (skills, tools, etc.). These resources will serve as the central focus of the educational intervention, and may undergo appropriate adjustments established during the co-creation sessions.
  2. MOOC acceptability and effectiveness: evaluation of the MOOC in terms of effectiveness (level of Health Literacy, Digital Health Literacy, and knowledge acquired) and acceptability (usability, areas for improvement, etc.)

SUMMARY:
The goal of this clinical trial is to promote Person-Centered Care and improve Health Literacy and Digital Health Literacy in women with breast cancer through the development of a Massive Open Online Course (MOOC) co-created with women with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult women ( ≥18 years old)
* Speak Spanish
* With internet at home or smartphone
* Currently have or have had breast cancer (currently disease-free)
* Families/caregivers of women with breast cancer and healthcare professionals involved in breast cancer management (oncologists, gynaecologists, nurses, psycho-oncologists, etc.)

Exclusion Criteria:

* No exclusion criteria were applied based on diagnosis date, current or past treatment, nationality, Health Literacy and Digital Health Literacy level and knowledge about Person-Centred Care or breast cancer.
* In the assessment of the MOOC's acceptability and effectiveness, participants involved in co-creating the MOOC will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Digital Health Literacy | Immediately after the intervention
  Digital Health Literacy through the eHealth Literacy Scale (eHEALS). It is an 8-item scale that uses a 5-point Likert scale to answer each question with response options ranging from "strongly agree" to "strongly disagree", resulting in a total score ranging from 8 to 40.
Health Literacy | Immediately after the intervention
  Health Literacy through the Health Literacy Survey European Questionnaire-16 items (HLS-EU-Q16). It is an abbreviated version of the Health Literacy Survey European Questionnaire (HLS-EU-Q) and consists of 16 items, with each question answered by choosing one response from the options: 'very difficult', 'fairly difficult', 'fairly easy', and 'very easy' giving a total score from 16 to 64.
Knowledge acquired | Immediately after the intervention
  Knowledge acquired before study each unit of the MOOC using a scale designed specifically for the study and in accordance with the content of each unit
Acceptability of MOOC | Immediately after the intervention
  Acceptability (usability, areas for improvement, etc.) of the MOOC using a scale designed specifically for the study, adhering to the methodology of the technology acceptance model (TAM)

CONTACTS AND LOCATIONS:
Locations (1):
- Servicio de Evaluación del Servicio Canario de la Salud, Santa Cruz de Tenerife, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvarez-Perez Y, Duarte-Diaz A, Toledo-Chavarri A, Abt-Sacks A, Ramos-Garcia V, Torres-Castano A, Rivero-Santana A, Perestelo-Perez L. Digital Health Literacy and Person-Centred Care: Co-Creation of a Massive Open Online Course for Women with Breast Cancer. Int J Environ Res Public Health. 2023 Feb 22;20(5):3922. doi: 10.3390/ijerph20053922. PMID 36900935